CLINICAL TRIAL: NCT04739566
Title: Dabrafenib and Trametinib Combination as a Neoadjuvant Strategy in BRAF-positive Anaplastic Thyroid Cancer (ANAPLAST-NEO)
Brief Title: Dabrafenib and Trametinib Combination as a Neoadjuvant Strategy in BRAF-positive Anaplastic Thyroid Cancer
Acronym: ANAPLAST-NEO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2021-01-29; First posted 2021-02-04 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Gland Anaplastic Carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (dabrafenib, trametinib) (Experimental): Patients receive dabrafenib 150 mg orally (PO) twice daily, trametinib 2mg PO once daily for 3 months
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Given PO twice daily
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
Drug: Trametinib — Given PO once daily
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
The aim of the study was to evaluate the effectiveness of combination therapy with dabrafenib and trametinib (anti-BRAF and anti-MEK inhibitors) in the neoadjuvant treatment of BRAF-positive anaplastic thyroid cancer. The prognosis in patients with ATC is poor due to the rapid and invasive tumor growth and the rapid development of metastases.

Dabrafenib is an antineoplastic agent, a selective RAF kinase inhibitor that competes with ATP. Oncogenic substitutions of the amino acid valine at position 600 (V600) BRAF lead to constitutive activation of the RAS / RAF / MEK / ERK pathway and stimulation of tumor cell growth.

Trametinib is a reversible, highly selective, allosteric inhibitor of the activation of mitogen-activated, extracellular signal-regulated kinases 1 (MEK1) and 2 (MEK2).

Dabrafenib and trametinib inhibit two kinases in the signaling pathway, BRAF, and MEK. The combination of the two drugs provides effective inhibition of proliferative signal conduction.

The investigators hypothesize that the combination treatment with these two drugs - dabrafenib and trametinib - can improve the response rate in the neoadjuvant mode in ATC without significant regimen-limiting toxicity and with better follow-up locoregional control.

DETAILED DESCRIPTION:
Primary endpoint

1. Objective Response Ratio (ORR) Evaluate the effectiveness of the combination of dabrafenib and trametinib using an objective response rate (ORR) for BRAF-mutated anaplastic thyroid cancer in neoadjuvant mode 7, 14, 28 days, 12, and 24 weeks after the start of treatment. Includes patients with a confirmed partial (PR) and complete response (CR) as the best response according to RECIST v 1.1.
2. Number of R0 resections after 3 months of neoadjuvant combination therapy with anti-BRAF and MEK inhibitors.

Comparison of the proportion of complete surgical resection (surgical resection R0 or R1) with historical controls of 5%. The R0 / R1 ratio will be determined by the proportion of patients who successfully undergo thyroidectomy with clear (R0) or microscopically positive (R1) resection margins.

Secondary endpoints

1. Safety Profile (Number / Severity of Serious Adverse Events, SAEs) Number of serious adverse events classified by severity as assessed by CTCAE v 5.0
2. Percentage of patients who received a complete response 3 months after the first dose of treatment.
3. Health-related quality of life Changes in health-related quality of life will be measured using the European Quality of Life Assessment Questionnaire (EQ-5D). The EQ-5D consists of a description and a health assessment. The health description consists of five dimensions (mobility, self-care, normal activities, pain/discomfort, and anxiety/depression), with each dimension identifying five levels of severity [best (1) - worst (5)]. Health assessment is assessed using a visual analog scale ([worse (0) - better (100)].
4. Progression-Free Survival (PFS) Median progression-free survival (mPFS) is defined as the time from the date of inclusion to the date of the first documented progression of disease or death from any cause, whichever occurs first. PFS will be determined based on the tumor score (RECIST criteria version 1.1).
5. Overall Survival (OS) Median overall survival (mOS) at 12, 24, 36, 48, and 60 months are calculated as the time from the date of inclusion to the date of death for any reason at the specific time points.

OUTLINE:

Patients receive dabrafenib orally (PO) twice daily (BID) and trametinib PO once daily (QD) for 3 months in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

After completion of study treatment, patients are followed up every 3 months during years 1-2, every 6 months during years 3-4, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years of age.
2. Willingness to participate in the study by signing an informed consent form approved by the ethics committee of the KVMT named after N.I. Pirogov St. Petersburg State University.
3. ECOG status 0 or 1 or 2. The ECOG assessment must be completed within 7 days prior to the distribution date.
4. Measurable disease according to RECIST 1.1, as defined by the investigator.
5. Patients with a histologically confirmed disease (according to the pathologist's report) that meets one of the following criteria (according to 2010 WHO classification):

   BRAF - positive anaplastic thyroid cancer, determined by immunohistochemistry for the presence of the BRAF V600E mutation in tumor tissue, genetic/molecular testing of the tumor, or by liquid biopsy of circulating DNA to determine the presence of the BRAF V600E mutation (if the histological examination is not possible). The primary tumor may or may not be resectable, but the risk of aerodigestive compression or bleeding should be excluded.
6. Weight over 30 kg.
7. Ability to swallow tablets/capsules or gastrostomy.
8. The absence of metastases in the brain.
9. Normal organ and bone marrow function as defined below (obtained = <30 days prior to study entry):

   * Hemoglobin ≥ 9.0 g / dL.
   * Absolute neutrophil count (ANC)> 1500 per mm.
   * Platelet count ≥ 100,000 per mm.
   * Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN) if liver metastases are absent, in which case it should be ≤ 2X ULN. This does not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, which is predominantly unconjugated in the absence of hemolysis or liver pathology); however, they will only be admitted after consulting their doctor.
   * Aspartate transaminase (AST) (SGOT) / alanine aminotransferase (ALT) (SGPT) ≤ 2.5x the institutional upper limit of normal, unless liver metastases are present, in which case it should be ≤ 5x ULN.
   * Measured creatinine clearance (CL)> 40 ml/min or Estimated creatinine clearance> 40 ml/min using the Cockcroft-Gault formula (Cockcroft and Gault, 1976) or 24-hour urine collection to determine creatinine clearance.
   * Albumin> = 2.5 mg / dL (received = <30 days prior to registration)
   * International normalized ratio (INR) or prothrombin time (PT) = <1.5 X ULN if the subject is not receiving anticoagulant therapy while PT or partial thromboplastin time (PTT) is within the therapeutic range of the intended use of anticoagulants
   * Activated partial thromboplastin time (APTT) = <1.5 x ULN if the subject is not receiving anticoagulant therapy while the PT or PTT is within the therapeutic range of the intended use of anticoagulants
10. Adequately controlled blood pressure with or without antihypertensive drugs, defined as blood pressure (BP) <150/90 mm Hg. Art.
11. Subjects should be prepared to undergo tumor biopsy before and after dabrafenib/trametinib therapy if a biopsy is impractical or not safe in the judgment of the treating physician. Subjects should be prepared for surgery if their tumor becomes surgically resectable. Research Subjects reserve the right to refuse any research intervention.
12. Female subjects of childbearing age (not surgically sterile or at least 2 years postmenopausal) must present a negative pregnancy test at screening and use a medically accepted double-barrier method of contraception (such as a spermicide condom + IUD or cervical caps) ... In addition, they must agree to continue using this double-barrier method for the duration of the study and for 4 months after the end of study participation. Women will be considered postmenopausal if they have had amenorrhea within 12 months without an alternative medical cause. The following age requirements apply:

    1. Women younger than 50 are considered postmenopausal if they have had amenorrhea for 12 months or more after stopping treatment with exogenous hormones, and if they have postmenopausal levels of luteinizing hormone and follicle-stimulating hormone or have undergone surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women over 50 years of age will be considered postmenopausal if they have had amenorrhea for 12 months or more after stopping all exogenous hormonal drugs with last menstrual period> 1 year ago, had menopause caused by chemotherapy with last menstrual period> 1 year ago, or have undergone surgery sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Men must agree to abstain from sexual intercourse with a female partner or agree to use a double-barrier method of contraception (for example, a spermicide condom, in addition to the fact that their female partner is using some form of contraception, such as an intrauterine device (IUD) or cervical caps), at the time of the study and for 4 months after the end of participation in the study, and refrain from donating sperm during this period.
14. Patient willingness and ability to adhere to protocol throughout the study, including undergoing treatment, and availability for scheduled visits and examinations, including follow-up.

Exclusion Criteria:

1. Concurrent participation in another clinical trial unless it is an observational (non-interventional) clinical trial or during the follow-up period of an interventional trial.
2. Taking any type of low molecular weight kinase inhibitor (including the investigational kinase inhibitor) for 2 weeks or 5 half-lives of the agent, whichever is greater.
3. Receiving any type of anticancer drugs (including investigational) or systemic chemotherapy within 2 weeks before starting treatment.
4. The presence of distant metastases (for example, to the brain, lungs).
5. Subject has an uncontrolled, serious underlying medical condition or recent illness, including but not limited to the following conditions:

   A) Cardiovascular diseases:
   * Congestive heart failure, grade 3 or 4 as defined by the New York Heart Association, unstable angina, and severe cardiac arrhythmias.
   * Uncontrolled hypertension, defined as sustained blood pressure> 150 mm Hg. Systolic or diastolic> 100 mmHg
   * Stroke, including transient ischemic attack (TIA), myocardial infarction, other ischemic event or thromboembolic events such as deep vein thrombosis (DVT) and pulmonary embolism) within 6 months prior to inclusion. Subjects with a later diagnosis of DVT are eligible if they are stable, asymptomatic, and have received LMWH for at least 6 weeks prior to study treatment.

   B) Gastrointestinal disorders (eg malabsorption syndrome or gastric outlet obstruction), including those associated with a high risk of perforation or fistula formation:
   * Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreas or bile ducts, or obstruction of the gastric outlet.
   * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months prior to inclusion. Note: Complete healing of the intra-abdominal abscess must be confirmed before starting treatment.

   C) Clinically significant vomiting or hemoptysis> 0.5 teaspoons (> 2.5 ml) of red blood or another significant bleeding in history within 3 months prior to treatment.

   D) Interstitial lung lesions or known manifestations of the endobronchial disease.

   F) Lesions invading the main pulmonary blood vessels.

   F) Other clinically significant disorders such as:
   * An active infection requiring systemic treatment, infection with human immunodeficiency virus or disease associated with acquired immunodeficiency syndrome, or chronic infection with hepatitis B or C.
   * Serious non-healing wound / ulcer / bone fracture.
   * Moderate or severe liver failure (Child-Pugh B or C).
   * The need for hemodialysis or peritoneal dialysis.
   * Uncontrolled diabetes mellitus.
   * History of solid organ transplantation.
6. Major surgery (such as gastrointestinal surgery and removal or biopsy of brain metastases) within 8 weeks prior to inclusion. Complete wound healing following major surgery should occur 4 weeks before the study treatment, and after minor surgery (eg, simple excision, tooth extraction) at least 10 days before the study treatment. Patients with clinically significant ongoing complications from prior surgery are not eligible.
7. Adjusted QT interval calculated by Fridericia formula (QTcf)> 500 ms for 28 days prior to study treatment.

   Note: If a single ECG displays a QTCf with an absolute value> 500 ms, two additional ECGs at approximately 3 min intervals must be performed within 30 minutes of the initial ECG, and the average of these three consecutive results will be used to assess eligibility for study participation.
8. Pregnant (test must be done no later than 7 days before the start of the study) or nursing mothers.
9. Received any live vaccine = <30 days prior to study initiation.
10. Inability to swallow tablets/capsules and lack of gastrostomy.
11. Previously identified allergy or hypersensitivity to the components of the investigational dosage forms.
12. Presence of previously diagnosed retinal vein occlusion, central serous retinopathy, uncontrolled glaucoma, or ocular hypertension.
13. Diagnosis of another malignant neoplasm within 3 years prior to study treatment, with the exception of superficial skin cancer or localized low-grade tumors that are considered cured and untreated by systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Prior to study completion, average 3 years
  Evaluate the effectiveness of the combination of dabrafenib and trametinib using an overall response rate (ORR) for BRAF-mutated anaplastic thyroid cancer in neoadjuvant mode 7, 14, 28 days, 12 and 24 weeks after the start of treatment. Includes patients with a confirmed partial (PR) and complete response (CR) as the best response according to RECIST v 1.1.
  ORR will be calculated as the number of patients with an observed response divided by the number of patients included in the study. A two-sided confidence interval will be calculated at 80% (in accordance with the specified α) and 95% (for comparison with the literature).
Number of R0 resections after 3 months of neoadjuvant combination therapy with anti-BRAF and MEK inhibitors. | 3 months
  Comparison of the proportion of complete surgical resection (surgical resection R0 or R1) with historical controls of 5 percent. The R0 / R1 ratio will be determined by the proportion of patients who successfully undergo thyroidectomy with clear (R0) or microscopically positive (R1) resection margins.

SECONDARY OUTCOMES:
Safety Profile (Number / Severity of Serious Adverse Events, SAEs) | SAEs will be reported in the clinical trial within 6 months of the end of the study.
  Number of serious adverse events classified by severity as assessed by CTCAE v 5.0
Percentage of patients who received a complete response 3 months after the first dose of treatment. | 3 months
  Percentage of patients who received a complete response 3 months after the first dose of treatment.
Health-related quality of life | up to 60 months
  Changes in health-related quality of life will be measured using the European Quality of Life Assessment Questionnaire (EQ-5D). The EQ-5D consists of a description and a health assessment. The health description consists of five dimensions (mobility, self-care, normal activities, pain / discomfort, and anxiety / depression), with each dimension identifying five levels of severity [best (1) - worst (5)]. Health assessment is assessed using a visual analogue scale ([worse (0) - better (100)].
Progression-Free Survival (PFS) | from date of enrollment to date of first documented progression, date of death from any cause, or patient failure, whichever is earlier, up to 60 months
  Median progression-free survival (mPFS) is defined as the time from the date of inclusion to the date of the first documented progression of disease or death from any cause, whichever occurs first. PFS will be determined based on the tumor score (RECIST criteria version 1.1).
Overall Survival (OS) | from date of enrollment to date of death from any cause or patient failure, whichever comes first, estimated up to 60 months
  Median overall survival (mOS) at 12, 24, 36, 48 and 60 months is calculated as the time from the date of inclusion to the date of death for any reason at the specific time points.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Mikheeva, M.D., Ph.D., Principal Investigator — Saint-Petersburg State University (SPSU) N.I.Pirogov Clinic of High Medical Technologies
Locations (1):
- Saint-Petersburg State University (SPSU) N.I.Pirogov Clinic of High Medical Technologies, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No